CLINICAL TRIAL: NCT04924374
Title: Microbiota Transplant in Advanced Lung Cancer Treated With Immunotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MORELIA
Record Dates: First submitted 2021-05-07; First posted 2021-06-14 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
Keywords: Oncology; Fecal Microbiota Transplantation; Metabolomics; Chemotherapy; Lung Cancer; Immunotherapy; Immunosenescence; Microbiota; Metagenomics; Metaproteomics
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — atezolizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti PD1 therapy plus Microbiota Transplant (Experimental): Active arm: Pooled fecal microbiota capsules of 1 donor selected based on their fecal abundance in Faecalibacterium prausnitzii, Bifidobacterium longum, Akkermansia muciniphila and Fusobacterium spp. after screening and metagenomic analysis of 10 donors with high-fiber diets (>30g/day).
  anti PD1 therapy every 2-3 weeks
  Interventions: Dietary Supplement: Microbiota Transplant plus anti PD1 therapy
- anti PD1 therapy (Active Comparator): Control arm: no intervention before anti PD1 therapy
  Interventions: Drug: anti PD1 therapy

INTERVENTIONS:
Dietary Supplement: Microbiota Transplant plus anti PD1 therapy — Pooled fecal microbiota capsules of 1 donor selected based on their fecal abundance in Faecalibacterium prausnitzii, Bifidobacterium longum, Akkermansia muciniphila and Fusobacterium spp. after screening and metagenomic analysis of 10 donors with high-fiber diets (>30g/day).
  anti PD1 therapy every 2-3 weeks
  Other Names: anti PD1 therapy Pembrolizumab, Nivolizumab, Atezolizumab
  Arms: anti PD1 therapy plus Microbiota Transplant
Drug: anti PD1 therapy — anti PD1 therapy every 2-3 weeks
  Other Names: Pembrolizumab, Nivolizumab, Atezolizumab
  Arms: anti PD1 therapy

SUMMARY:
The gut microbiota can modulate the effectiveness of cancer therapies, especially immunotherapy. Manipulating the microbial populations in patients with advanced lung cancer through fecal microbiota transplantation from healthy individuals or from long-term survivors to advanced lung cancer will enhance the efficacy of immunotherapy.

DETAILED DESCRIPTION:
Lung cancer is a leading cause of mortality worldwide, and its treatment and prognosis are being revolutionized by immunotherapy. The gut microbiome has been shown able to modulate the antitumor efficacy of immunotherapeutic agents in pre-clinical models, demonstrating that patients can be stratified into responders and nonresponders to immunotherapy on the basis of their microbiota composition. Fecal microbiota transplants have demonstrated to improve the efficacy of immunotherapy in animal models. In this study, investigators will include 20 stage III/V non-small cell lung cancer naïve for PD/PD L-1 inhibitors that require treatment in monotherapy or combined with chemotherapy as consolidation strategy after concurrent chemotherapy and radiotherapy (stage III), upfront treatment (stage IV patients with PDL1 status > 50%) or as second line strategy for those patients with advanced disease who progressed to chemotherapy alone. The participants will be randomized to receive either fecal microbiota capsules from 3 donors selected based on the fecal abundance of bacterial taxa shown to correlate with a greater response to immunotherapy or not, in combination with the PDL/PDL1 agent. The primary outcome will be safety. The secondary outcomes will be treatment response (iRECIST criteria). Investigators will also examine engraftment of donor's microbiota on host microbiota using Illumina DNA shotgun sequencing, changes in the bacterial metabolism using metaproteomics, and in the plasma metabolite fingerprint by untargeted mass spectrometry in bacterial and plasma samples, and changes in peripheral immune cells subpopulations and antitumoral immunity. MORELIA could improve the prognosis of a lung cancer in a subset of patients with limited therapeutic options and inform on how to exploit host-microbiota interactions with tailored fecal microbiota transplantation to boost the clinical response to immunotherapy in advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent
2. Age >18 years.
3. Diagnosis of unresectable stage III non-small cell cancer histologically or citologically confirmed.
4. Eastern Cooperative Oncology Group (ECOG) Score ≤1
5. Disease able to be monitored using the RECIST v.1.1. criteria (lesions treated with radiotherapy can be defined as target lesions if the progression has been documented).
6. At least 3 weeks since the last treatment for cancer, including chemotherapy and radiotherapy when combined in stage III patients, and recovery ≤1 from any adverse event related with previous treatment for cancer, excluding sensorial neuropathy, anemia, asthenia, hair loss, all grade ≤2), according to the National Cancer Institute (CTCAE del NCI, v.5) definitions
7. Adequate bone marrow, renal, liver and metabolic parameters (evaluated at least 7 days prior the inclusion in the study:

   * Platelet count ≥100 x 109/l, hemoglobin ≥9 g/dl and absolute neutrophil count ≥1,000 x 109/l.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times the upper limit of normality, independently of the presence of liver metastases.
   * Alkaline phosphatase ≤ 2,5 times the upper limit of normality.
   * Total bilirubin ≤1,5 times the upper limit of normality o direct bilirubin below the upper level of normality.
   * INR<1,5, except if concomitant oral anticoagulation
   * Estimated glomerular filtration rate ≥30 ml/minute using the EPI equation
   * Albumin ≥3 g/dl without previous parenteral albumin treatment.
8. All men and women with childbearing potential must accept the use of highly efficacious contraceptive methods during the study.

Exclusion Criteria:

1. Active of untreated central nervous system (CNS) involvement. Treated CNS metastases must be radiologically stable (defined as the absence of CNS progression during at least 3 weeks from the first CNS imaging after radiotherapy to the CNS imaging prior the screening visit. Participants will not be included in the presence of any neurological sign or symptom secondary to CNS metastases or radiotherapy. Any treatment with steroids must have been completed at least 14 days before the first study intervention.
2. Prior use of immunotherapy of immunomodulatory treatment for non-small cell lung cancer, either in combination or in monotherapy, at any stage of the disease.
3. Radiotherapy in >35% the bone marrow.
4. Prior bone marrow or cell-stem transplant.
5. Treatment with immunoestimulatory agents, including interferons or interleukin-2 before 4 weeks or 5 drug half-lives (whichever longer) before the randomization.
6. Prior neoplasia, with the exception of skin basocelular carcinoma, superficial bladder carcinoma, squamous cell skin carcinoma, cervix high degree intrasquamous lesion. Those patients with prior neoplasia free of recurrence during at least 2 years are eligible.
7. Severe infections four weeks before the screening, including hospitalization due to any infection, bacteremia or severe pneumonia.
8. Rectal colonization by vancomycin resistant enterococci
9. Overt immunodeficiency, including systemic treatment with steroids at >10 mg of prednisone/day (or its equivalent) or other immunosuppressive agents during the 14 days before the first study intervention.
10. Moderates-severe mucositis , GI symptoms
11. Dysphagia, history of aspirative pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Measure of safety | 27 weeks
  The safety variables (vital signs, physical examinations, symptoms, laboratory test results and the occurrence of adverse events) will be assessed at each visit. The incidence of adverse events will be categorized by severity and related to the time of occurrence. Changes in physical examinations, changes in laboratory test results (hematology, biochemistry and urinalysis tests) from screening period, and change of vital signs will be summarized and analyzed by the descriptive statistics. Adverse events will be defined according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria. v5.0

SECONDARY OUTCOMES:
Measure of Efficacy | 27 weeks
  Immunotherapy Response Evaluation Criteria in Solid Tumors-iRECIST

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided